CLINICAL TRIAL: NCT03940014
Title: Pulmonary Arteriovenous Malformations (PAVMs) in Hereditary Haemorrhagic Telangiectasia (HHT): Correlations Between Computed Tomography Findings and Cerebral Complications
Brief Title: Pulmonary Arteriovenous Malformations (PAVMs) in Hereditary Haemorrhagic Telangiectasia (HHT)
Acronym: PAVM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: PAVM
Record Dates: First submitted 2019-05-02; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Hereditary Haemorrhagic Telangiectasia; Pulmonary Arteriovenous Malformation; Cerebral Disorder
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Pulmonary Arteriovenous Fistulas

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary arteriovenous malformations: Patients with hereditary haemorrhagic telangiectasia (HHT)-related Pulmonary Arteriovenous Malformations (PAVMs). For all patients, the final diagnosis of certain HHT the diagnosis can be made depending on the presence of four criteria known as the Curaçao criteria: 1) Spontaneous recurrent epistaxis 2) Multiple telangiectasias in typical locations 3) Proven visceral Arteriovenous Malformations (AVM) (lung, liver, brain, spine) 4) First-degree family member with HHT. If conditions three or four are met, a patient has "definite HHT", while condition two is considered as "possible HHT". All patients had a molecular diagnosis and all follow-up clinical assessments were available in the database.
  Interventions: Other: Data collection from standard follow up

INTERVENTIONS:
Other: Data collection from standard follow up — Annual clinical consultation with an Hereditary Haemorrhagic Telangiectasia (HHT) specialist and/or pneumologist and organ specialists when necessary (such as hepatologists, cardiologists and neurologists).
  Explorations (contrast echography, chest Computed Tomography and treatments performed according to international guidelines.
  TransCatheter Embolotherapy for each treatable Pulmonary Arteriovenous Malformations (PAVMs) and follow-up every 3 years.
  Chest Computed Tomography (CT) every 6-12 months.

SUMMARY:
Computed tomography (CT) is the modality of choice to characterize pulmonary arteriovenous malformations (PAVMs) in patients with hereditary haemorrhagic telangiectasia (HHT). The objective of this study was to determine if CT findings were associated with frequency of brain abscess and ischaemic stroke.

This retrospective study included patients with HHT-related PAVMs. CT results, PAVM presentation (unique, multiple, disseminated or diffuse), the number of PAVMs and the largest feeding artery size, were correlated to prevalence of ischaemic stroke and brain abscess.

ELIGIBILITY:
Inclusion Criteria:

* Hereditary Haemorrhagic Telangiectasia (HHT) diagnosis
* Pulmonary Arteriovenous Malformations (PAVMs) related with HHT

Exclusion Criteria:

* Clinical follow-up not available in the database

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hereditary Haemorrhagic Telangiectasia (HHT) Patients who had a molecular diagnosis and all follow-up clinical assessments available in the database.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Yearly change in chest Computed Tomography (CT) results in patients with Hereditary Haemorrhagic Telangiectasia (HHT). | Every year for 10 years
  The presence of pulmonary arteriovenous malformations (PAVMs) (unique, multiple, disseminated or diffuse, the number of PAVMs and the largest feeding artery size) upon examination by CT could be correlated to the frequency of brain abscess and ischemic stroke in patients with hereditary haemorrhagic telangiectasia (HHT). These patients underwent a yearly CT scan to check for PAVM presence.

CONTACTS AND LOCATIONS:
Overall Officials: Salim Si-Mohamed, MD, Principal Investigator — Hospices Civils de Lyon (Hôpital cardiologique Louis Pradel)